CLINICAL TRIAL: NCT06838546
Title: A Multicenter, Open Phase IIb Clinical Study to Evaluate the Efficacy and Safety of B1962 Injection in the Treatment of Advanced Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tasly Biopharmaceuticals Co., Ltd. (Industry)
Collaborators: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSL-B1962-03
Record Dates: First submitted 2025-02-17; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Advanced Colorectal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- B1962 (Experimental): advanced colorectal cancer
  Interventions: Drug: B1962

INTERVENTIONS:
Drug: B1962 — B1962 has higher VEGF anti angiogenic activity than its competitors. Phase I clinical trials have shown that B1962 has excellent safety and promising therapeutic effects. Large scale clinical studies may achieve better therapeutic effects than similar competitors targeting the same target
  Other Names: B1962 is a PD-L1/VEGF bispecific antibody fusion protein.

SUMMARY:
This is a multicenter, randomized, open-label, two-stage Phase IIb clinical study to evaluate the efficacy and safety of B1962 in the treatment of advanced colorectal cancer.

The subjects were patients with distant metastasis or unresectable locally advanced colorectal cancer who had previously failed oxaliplatin, irinotecan, fluorouracil-based drugs therapy containing disease progression or intolerable toxic side effects.

Two dose groups were investigated:

Dose group 1: B1962 35 mg/kg, intravenous infusion, Q2W, Dose group 2: B1962 45 mg/kg, intravenous infusion, Q2W.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for enrollment in this study:

1. Voluntary participation in the study and provision of signed and dated informed consent;
2. Aged 18 to 75 years (inclusive) at the time of signing informed consent;
3. Patients with distant metastasis or unresectable locally advanced colorectal cancer who have disease progression or intolerable toxicities after previous standard treatment must include oxaliplatin, irinotecan and fluorouracil-based drugs in previous standard treatment regimen;
4. Histologically or cytopathologically confirmed adenocarcinoma of the colon or rectum, including adenocarcinoma of the appendix;
5. Willingness to comply with protocol-specified visits, study treatment, laboratory tests, and other study-related procedures and requirements;
6. Eastern Cooperative Oncology Group (ECOG) performance score 0-1;
7. Expected survival time of more than 3 months;
8. Presence of at least one measurable lesion (non-radiation field) confirmed by CT or MRI that meets RECIST v1.1 criteria;
9. Adequate organ and bone marrow function:

   Hematologic system (no transfusion, no G-CSF use, no medication correction within 2 weeks prior to screening): absolute neutrophil count (ANC) ≥ 1.5 × 10 9/L, platelets (PLT) ≥ 75 × 10 9/L, hemoglobin (Hb) ≥ 90 g/L; Liver function: total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN), alanine aminotransferase (ALT) ≤ 3.0 × ULN, aspartate aminotransferase (AST) ≤ 3.0 × ULN; for patients with liver metastasis: ALT ≤ 5.0 × ULN, AST ≤ 5.0 × ULN; albumin ≥ 30 g/L; Renal function: creatinine within normal range, or creatinine clearance (Ccr) ≥ 60 mL/min (calculated according to Cockcroft-Gault formula); Cockcroft-Gault formula is: Ccr (ml/min) = [(140-age) × weight (kg)× F]/[serum creatinine (mg/dl) × 72] (F = 1 for males and 0.85 for females) Urine protein was qualitatively 0, ±, or < 0.5 g/24 hours. All patients with urine protein(±) in urinalysis must have a 24-hour urine collection and must demonstrate urine protein < 0.5 g/24 hours.

   Coagulation: prothrombin time (PT) ≤ 1.5 × ULN or international normalized ratio (INR) ≤ 1.5 × ULN, and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN;
10. Fertile subjects agree to use highly effective contraception from signing the ICF and to avoid pregnancy during the study and for 3 months after the last dose (male or female subjects)

    * Females of childbearing potential must be non-lactating and agree to use highly effective contraception from signing the ICF, and must practice contraception during the study and for 3 months after the last dose; blood pregnancy results (human chorionic gonadotropin hCG) must be negative within 7 days prior to enrollment;
    * Females of non-childbearing potential (ie, physiologically incapable of becoming pregnant), including those who have been surgically sterilized (having undergone bilateral oophorectomy, bilateral tubal ligation, or hysterectomy), or who have been postmenopausal for ≥ 12 months prior to Screening (amenorrhea not due to treatment).

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study:

1. Prior therapy targeting PD- (L) 1 and VEGF/VEGFR, including concurrent use of anti-PD-1/PD-L1 monoclonal antibody in combination with drugs targeting VEGF/VEGFR, or anti-PD-1/VEGF or anti-PD-L1/VEGF bispecific antibodies or bispecific fusion proteins, or sequential use of anti-PD-1/PD-L1 monoclonal antibody and drugs targeting VEGF/VEGFR;
2. Received the last systemic anti-tumor treatment (biological agent therapy, etc.) within 4 weeks before the first dose, hormone anti-tumor treatment within 2 weeks before the first dose, non-specific immunomodulatory treatment (such as interleukin, interferon, thymosin, thalidomide, tumor necrosis factor, etc.) within 2 weeks before the first dose, and received Chinese herbal medicine or Chinese patent medicine with anti-tumor indications within 1 week before the first dose;
3. Received systemic anti-tumor therapy in other clinical studies within 4 weeks prior to the first dose;
4. Radiotherapy or surgery within 4 weeks prior to the first dose and diagnostic biopsy within 7 days prior to the first dose;
5. Patients who have received live or attenuated vaccines within 4 weeks before screening or plan to receive live or attenuated vaccines during the study;
6. Known hypersensitivity to the study drug or any of its components, or previous severe hypersensitivity to macromolecular protein preparations/monoclonal antibodies or bispecific antibodies;
7. Adverse reactions from prior anticancer therapy that have not recovered to NCI-CTCAE v5.0 grade ≤ 1 (except alopecia, etc. for which the investigator considers there is no safety risk);
8. Prior therapy with ≥ Grade 1 proteinuria, or prior bleeding event ≥ Grade 2 related to drugs targeting VEGF/VEGFR, or prior therapy with ≥ Grade 3 hypertension or ≥ Grade 3 immune-related adverse event.
9. Known brain and/or leptomeningeal metastases;
10. Patients with pleural effusion, pericardial effusion or peritoneal effusion accompanied by clinical symptoms, or pleural effusion, pericardial effusion or ascites that cannot be controlled by treatment of primary disease, anti-tuberculosis, anti-infection, diuretics or requires repeated drainage once every 3 weeks or more frequently;
11. Complete or incomplete bowel obstruction or risk of bowel obstruction reported on imaging studies, presence of intra-abdominal abscess, or history of inflammatory bowel disease (eg, Crohn 's disease, ulcerative colitis);
12. Screening imaging showed tumor encasing vital vessels or obvious necrosis and cavity, and the investigator judged that entering the study would cause bleeding risk, or tumor invading vital organs (such as heart and pericardium, trachea, esophagus) or risk of esophagotracheal fistula or esophagopleural fistula , ulcerated colorectal cancer or tumor infiltrating the full thickness of intestinal wall, or other lesions involving the gastrointestinal tract with bleeding or gastrointestinal fistula and gastrointestinal perforation risk;
13. Known history of human immunodeficiency virus (HIV) infection (HIV 1/2 antibody positive) or acquired immunodeficiency syndrome-related diseases, or other immunodeficiency diseases;
14. Positive hepatitis B surface antigen (HBsAg), and HBV DNA higher than the upper limit of normal value of the detection unit; or positive hepatitis C antibody (HCV-Ab) and HCV-RNA quantification > the upper limit of normal value of the detection unit; or known active syphilis infection;
15. Fever of unknown origin > 38.5℃; or bacterial, viral, fungal infections and other pathogen infections (such as mycoplasma, parasites, etc.) requiring systemic treatment; or uncontrolled active infections such as tuberculosis;
16. History of significant cardiovascular disease, including but not limited to: malignant arrhythmia requiring clinical intervention; or acute coronary syndrome (myocardial infarction and angina pectoris) or coronary artery bypass grafting within 6 months before the first dose; or congestive heart failure meeting New York Heart Association (NYHA) functional class II or higher criteria; or left ventricular ejection fraction (LVEF) < 50%; poor compliance with standard treatment for hypertension or antihypertensive therapy; history of hypertensive crisis or hypertensive encephalopathy; major vascular disease (e.g., aortic aneurysm requiring surgery);
17. Patients suffering from coagulation disorders, bleeding disorders, or other bleeding risks judged by the investigator, such as skin wounds, surgical sites, wound sites, severe mucosal ulcers, fractures, intestinal fistulas without complete healing, or active gastric or duodenal ulcers, gastrointestinal bleeding, esophageal and gastric varices, gastrointestinal perforation within 6 months before the first dose;
18. Pulmonary hemorrhage/hemoptysis (daily bleeding/hemoptysis volume ≥ 2.5ml) within 4 weeks prior to the first dose of study drug;
19. Arterial or venous thrombosis, or stroke or transient ischemic attack within 6 months prior to the first dose of study drug;
20. Unstable anticoagulant or thrombolytic therapy within 14 days of the first dose of study drug;
21. Chronic treatment with aspirin (> 325 mg/day) or nonsteroidal anti-inflammatory drugs known to inhibit platelet function, or thienopyridines such as ticlopidine, clopidogrel, or phosphodiesterase inhibitors such as dipyridamole, cilostazol within 14 days of the first dose of study drug;
22. Diabetes mellitus and thyroid diseases not stably controlled by drug therapy, such as hyperthyroidism;
23. Current or past idiopathic pulmonary fibrosis or idiopathic pneumonia; current acute lung disease, interstitial lung disease or pneumonia, pulmonary fibrosis, etc.; severe dyspnea, pulmonary insufficiency or continuous oxygen inhalation for any reason;
24. Active autoimmune diseases or history of autoimmune diseases requiring systemic treatment within 2 years before screening, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vasculitis or glomerulonephritis;
25. Systemic corticosteroid therapy (prednisone > 10 mg/day or equivalent of the same class) or systemic therapy with other immunosuppressive agents within 14 days prior to the first dose of study drug;

Exceptions:

1. Topical, ocular, intra-articular, intranasal, or inhaled corticosteroid therapy with minimal systemic absorption;
2. Short-term (≤ 7 days) corticosteroid prophylaxis (eg, allergy to contrast agents) or treatment of non-autoimmune allergic diseases (eg, delayed hypersensitivity caused by contact allergens); 26.Prior organ or hematopoietic stem cell transplant; 27.History of other neoplasms within 5 years prior to screening, except cured cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, cervical carcinoma in situ, papillary thyroid carcinoma, who had undergone successful radical surgery; 28.History of substance abuse or mental disorder; Other serious systemic diseases or laboratory abnormalities or compliance problems or other reasons considered unsuitable for this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-24 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 24 months
  Proportion of patients who achieved complete response (CR) or partial response (PR) at two consecutive reviews ≥ 4 weeks apart.

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hanzhou, Hanzhou, China

IPD SHARING:
Plan to Share IPD: No